CLINICAL TRIAL: NCT04085757
Title: Determining the Optimal Time Interval Between Vaginal Dinoprostone Administration and Diagnostic Office Hysteroscopy in Nulliparous Women: A Randomized Double-Blind Trial
Brief Title: Optimal Timing of Dinoprostone Administration Prior to Office Hysteroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dinoprostone timing
Record Dates: First submitted 2019-09-07; First posted 2019-09-11 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Dinoprostone Timing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long interval dinoprostone (Experimental): A small envelope including two labeled plastic bags (A & B) (each bag containing either 1 dinoprostone tablet(3mg) or 1 identically appearing placebo tablet) will be packaged in sequentially numbered sealed envelopes. In long interval dinoprostone group, bag (A) contains dinoprostone tablet and bag (B) contains placebo tablet. After signing the informed consent, the sequentially numbered sealed envelopes will be opened (according to the sequence of attendance of the patient) by the study nurse. Tablets in bag (A) will be inserted 12 hours before office hysteroscopy and tablets in bag (B) will be inserted 3 hours before office hysteroscopy.
  Interventions: Drug: long interval dinoprostone
- short interval dinoprostone (Active Comparator): A small envelope including two labeled plastic bags (A& B) (each bag containing either 1 dinoprostone tablets(3 mg) or 1 identically appearing placebo tablet) will be packaged in sequentially numbered sealed envelopes. In short interval dinoprostone group, bag (A) contains placebo tablet and bag (B) contains dinoprostone tablet. After signing the informed consent, the sequentially numbered sealed envelopes will be opened (according to the sequence of attendance of the patient) by the study nurse. Tablets in bag (A) will be inserted 12 hours before office hysteroscopy and tablets in bag (B) will be inserted 3 hours before office hysteroscopy.
  Interventions: Drug: short interval dinoprostone

INTERVENTIONS:
Drug: long interval dinoprostone — A small envelope including two labeled plastic bags (A & B) (each bag containing either 1 dinoprostone tablet(3mg) or 1 identically appearing placebo tablet) will be packaged in sequentially numbered sealed envelopes. In long interval dinoprostone group, bag (A) contains dinoprostone tablet and bag (B) contains placebo tablet. After signing the informed consent, the sequentially numbered sealed envelopes will be opened (according to the sequence of attendance of the patient) by the study nurse. Tablets in bag (A) will be inserted 12 hours before office hysteroscopy and tablets in bag (B) will be inserted 3 hours before office hysteroscopy.
  Arms: long interval dinoprostone
Drug: short interval dinoprostone — A small envelope including two labeled plastic bags (A& B) (each bag containing either 1 dinoprostone tablet(3 mg) or 1 identically appearing placebo tablet) will be packaged in sequentially numbered sealed envelopes. In short interval dinoprostone group, bag (A) contains placebo tablet and bag (B) contains dinoprostone tablet. After signing the informed consent, the sequentially numbered sealed envelopes will be opened (according to the sequence of attendance of the patient) by the study nurse. Tablets in bag (A) will be inserted 12 hours before office hysteroscopy and tablets in bag (B) will be inserted 3 hours before office hysteroscopy.
  Arms: short interval dinoprostone

SUMMARY:
The aim of this study is to determine whether dinoprostone administered 10 hours before office hysteroscopy can relieve pain more effectively compared with dinoprostone administered 3 hours before office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous patients who have an indication for office hysteroscopy

Exclusion Criteria:

* Parous patients, menopausal patients and patients with cervical pathology, and previous cervical surgery will be excluded from the study. Moreover, patients with severe vaginal bleeding, allergy to dinoprostone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | intraoperative
  Intensity of pain by visual analog scale from 0(no pain) to 100 mm(worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - faculty of medicine Cairo university, Giza
  - Tertiary referral hospital, Giza

REFERENCES:
- [Derived] Rund NMA, El Shenoufy H, Islam BA, El Husseiny T, Nassar SA, Mohsen RA, Alaa D, Gad Allah SH, Bakry A, Refaat R, Gehad MA, Kotb MMM, Osman OM, Ashour ASA, Ali AS, Taher A, Kholaif K, Hashem AT, Elsallamy AAH, Nour DA, Dahab S, Talaat B, Almohammady M. Determining the Optimal Time Interval between Vaginal Dinoprostone Administration and Diagnostic Office Hysteroscopy in Nulliparous Women: A Randomized, Double-blind Trial. J Minim Invasive Gynecol. 2022 Jan;29(1):85-93. doi: 10.1016/j.jmig.2021.06.021. Epub 2021 Jul 1. PMID 34217851